CLINICAL TRIAL: NCT00002058
Title: A Randomized Controlled Prophylactic Study of Clofazimine To Prevent Mycobacterium Avium Complex Infection in HIV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 027A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-12

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Clofazimine; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Clofazimine

INTERVENTIONS:
Drug: Clofazimine

SUMMARY:
This study will examine the effectiveness of clofazimine in the prophylaxis of Mycobacterium avium complex infection in HIV infected individuals who are at risk to develop this untreatable opportunistic disease. In the absence of truly effective antiretroviral therapy, a potential mode of treatment of patients with HIV infection is to prevent the development of the life-threatening opportunistic infections. Current studies demonstrate a possible efficacy of clofazimine in the prophylaxis against Pneumocystis carinii pneumonia (PCP), the most common AIDS-defining opportunistic infection. Future studies will examine the potential for prophylaxis against the other opportunistic infections. This proposal hopes to define the role of prophylactic clofazimine in preventing the currently untreatable Mycobacterium avium complex infection. AMENDED: To include prophylaxis for Asymptomatic and ARC.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Pneumocystis prophylaxis.
* Antiretroviral therapy, or other experimental protocols.
* Antipyretics and analgesics as per the treating physician.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Unexplained fever.
* Night sweats.
* Unexplained anemia with hemoglobin < 10 g percent or hematocrit less than 30 percent.
* Hepatic transaminase elevations or total bilirubin values of > 3 times normal.
* Long-term (over 2 weeks) treatment with any drug with known significant anti-Mycobacterium avium complex (MAC) activity including isoniazid, ethambutol, rifampin, raffia, PAS, PZA, amikacin, streptomycin, ethionamide, viomycin, cycloserine, capreomycin, ciprofloxacin, imipenem, rifapentine, gentamicin, or penicillin.

Patients with the following are excluded:

* Known hypersensitivity to clofazimine.
* Mycobacterium avium complex (MAC) infection diagnosis at any site (except isolation from stool in asymptomatic patient).
* Any of the following symptoms at the time of study entry:
* Unexplained fever.
* Night sweats.
* Unexplained anemia with hemoglobin < 10 percent or hematocrit less than 30 percent.
* Hepatic transaminase elevations or total bilirubin values of > 3 times normal.
* Long-term (over 2 weeks) treatment with any drug with known significant anti-MAC activity.

Prior Medication:

Excluded:

* Long-term (over 2 weeks) treatment with any drug with known significant anti-Mycobacterium avium complex (MAC) activity including isoniazid, ethambutol, rifampin, raffia, PAS, PZA, amikacin, streptomycin, ethionamide, viomycin, cycloserine, capreomycin, ciprofloxacin, imipenem, rifapentine, gentamicin, or penicillin.

Group 1:

* AIDS patients with a first episode of Pneumocystis carinii pneumonia (PCP) within 2 to 4 months prior to study entry.
* Group 2:
* Patients with T4 counts < 100 cells/mm3, regardless of prior opportunistic infections or malignancies.
* Karnofsky = or > 70.
* All patients must sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Keith Med Group, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California

REFERENCES:
- [Background] Gustavson LE, Fukuda EK, Rubio FA, Dunton AW. A pilot study of the bioavailability and pharmacokinetics of 2',3'-dideoxycytidine in patients with AIDS or AIDS-related complex. J Acquir Immune Defic Syndr (1988). 1990;3(1):28-31. PMID 2152803
- [Background] Abrams DI, Mitchell TF, Child CC, Shiboski SC, Brosgart CL, Mass MM. Clofazimine as prophylaxis for disseminated Mycobacterium avium complex infection in AIDS. J Infect Dis. 1993 Jun;167(6):1459-63. doi: 10.1093/infdis/167.6.1459. PMID 8501340